CLINICAL TRIAL: NCT06856031
Title: A Retrospective Analysis on the Long-term Retention Rate and Influence Factors of Individualized Treatment of Vedolizumab in Patients With Ulcerative Colitis
Brief Title: the Long-term Retention Rate and Influence Factors of Individualized Treatment of Vedolizumab in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-204
Record Dates: First submitted 2025-02-10; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: IBD (Inflammatory Bowel Disease)
Keywords: Ulcerative colitis; vedolizumab; drug retention; influencing factors
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Optimized Treatment (OPT) — After induction therapy with intravenous vedolizumab (300 mg) at weeks 0, 2, and 6, PRO2 was assessed to determine the patient's response and an individualized treatment plan was formulated: vedolizumab was reinfused intravenously (300 mg) every 4 weeks if PRO2 was reduced by <50% from baseline or was still in the moderately-severe active phase of PRO2.

SUMMARY:
The drug retention rate of vedolizumab for ulcerative colitis decreases with time. This study analyzed the long-term drug retention rate and its influencing factors in patients with moderately to severely active ulcerative colitis treated with vedolizumab.

DETAILED DESCRIPTION:
Vedelizumab is a humanized monoclonal antibody that specifically recognizes α4β7 heterodimer, selectively blocks the interaction between mucosal addressin cell adhesion molecule-1 (MAdCAM-1) on intestinal blood vessels and α4β7 integrins on the surface of lymphocytes, inhibiting the migration of lymphocytes to the gastrointestinal mucosa and thus exerting anti-inflammatory effects. The regimen of vedolizumab therapy for the treatment of ulcerative colitis is intravenous vedolizumab (300 mg) at weeks 0, 2, and 6 for induction therapy, followed by intravenous vedolizumab (300 mg) every 8 weeks for maintenance therapy. This study analyzed the long-term drug retention rate and its influencing factors in moderately and severely active UC patients treated with VDZ, aiming to provide a more precise and personalized treatment plan for UC patients before initiating VDZ therapy, and to better predict drug efficacy as well as retention rate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with moderate to severe ulcerative colitis
2. Receiving treatment with vedolizumab

Exclusion Criteria:

1. Combination therapy with other biological agents, small molecule drugs, immunosuppressants or hormone therapy.
2. Combination of active tuberculosis, Clostridium difficile infection, cytomegalovirus infection, EBV infection, etc.
3. Combined with malignant tumors or autoimmune diseases (such as dry syndrome, systemic lupus erythematosus, rheumatoid arthritis, etc.).
4. Combined with serious cardiovascular and cerebrovascular diseases or liver and renal insufficiency.

   * Loss of visit or clinical data ≥30% during the follow-up period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inflammatory bowel disease (IBD) is a chronic inflammatory disease involving the digestive tract, including two clinical phenotypes: Crohn's disease (CD) and ulcerative colitis (UC).
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Drug retention rates analyzed at weeks 54 of vedolizumab treatment | at week 54
  the drug retention rate of vedolizumab
Drug retention rates analyzed at weeks 108 of vedolizumab treatment | at week 108
  the drug retention rate of vedolizumab

SECONDARY OUTCOMES:
Analyze the impact of baseline MES on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline MES between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
  The Mayo endoscopic score (MES) was used to assess the degree of intestinal inflammation, with a score of MES=0 defined as mucosal healing, MES=1 as mild, MES=2 as moderate, and MES=3 as severe.
Analyze the impact of baseline disease sites on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in disease sites between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
  Disease sites were categorized into proctitis (E1), left hemicolonitis (E2) and extensive colitis (E3) based on the Montreal UC phenotypic classification criteria.
Analyze the impact of baseline modified Mayo score on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in the baseline modified Mayo score between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment). The modified Mayo score was employed to assess UC disease activity. A modified Mayo score of ≤5 was defined as mild activity, 6-10 as moderate activity, and ≥11 as severe activity.
Analyze the impact of duration of disease on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in duration of disease (in years) between VDZ-continued group and VDZ-discontinued group.
Analyze the impact of baseline C-reactive protein in peripheral blood on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline C-reactive protein (mg/L) in peripheral blood between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analyze the impact of baseline erythrocyte sedimentation rate on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline erythrocyte sedimentation rate (mm/h) between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analyze the impact of baseline 25(OH) D in peripheral blood on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline 25(OH) D in peripheral blood (ng/mL) between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analyze the impact of baseline serum albumin in peripheral blood on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline serum albumin (g/L) in peripheral blood between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analysis of the impact of baseline absolute eosinophil count in peripheral blood on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline absolute eosinophil count in peripheral blood (×10^8) between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analysis of the impact of baseline hemoglobin in peripheral blood on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline hemoglobin in peripheral blood (g/L) between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analysis of the impact of baseline white blood cell count in peripheral blood on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline white blood cell count in peripheral blood (×10^9) between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analysis of the impact of baseline platelet count in peripheral blood on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline platelet count in peripheral blood (×10^9) between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment).
Analysis of the impact of baseline body mass index on VDZ drug retention rates | at week 54 and 108
  Analyze the difference in baseline body mass index between VDZ-continued group and VDZ-discontinued group (Baseline is defined as week 0 of VDZ treatment). Body Mass Index (BMI) is a numerical value derived from an individual's weight and height, calculated by dividing the weight in kilograms by the square of the height in meters (kg/m²). Baseline height (m) and weight (kg) of patients need be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No